CLINICAL TRIAL: NCT02980939
Title: The Role of Hydration on Exercise Performance - ODIN
Acronym: ODIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas, Fayetteville (Other)
Responsible Party: Principal Investigator, Stavros Kavouras, Associate Professor, University of Arkansas, Fayetteville
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 16-10-135
Record Dates: First submitted 2016-11-30; First posted 2016-12-02 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Dehydration
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Euhydration - no thirst (Placebo Comparator)
  Interventions: Other: iv fluid infusion
- Dehydration - no Thirst (Experimental)
  Interventions: Other: iv fluid infusion

INTERVENTIONS:
Other: iv fluid infusion — Intravenous isotonic saline infusion

SUMMARY:
During exercise in the heat, there is a need to replenish fluids in order to avoid dehydration and decrease the risk for heat illness. What drives this urge to drink is the thirst mechanism. Following ingestion of fluids, there is an inhibition of thirst before there is a replenishing of fluids. However, there is little scientific evidence of where thirst is inhibited, if this thirst inhibition is augmented by exercise and how thirst itself influence exercise performance. Further, during rehydration studies, it is very difficult to successfully blind a subject to their drinking/hydration protocol. Previous studies that have blinded a subject to their drinking have used various methods such as intravenous fluid administration and/or nasogastric tubes. Therefore, the purpose of this research is to examine the mechanistic roles thirst inhibition plays while exercising in the heat while undergoing intravenous fluid administration. Specific attention will be directed to the cardiovascular and thermoregulatory function of the individuals. All blood, cardiovascular, thermoregulatory, and perceptual measures are shown in the diagram below.

ELIGIBILITY:
Inclusion Criteria:

* Cycling Racing History category 3 or higher USA cycling certification
* maximal oxygen uptake >55 ml/kg/min

Exclusion Criteria:

* History of heat stroke
* Renal, cardiovascular, metabolic diseases
* Regular medication

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2016-11; Primary Completion 2017-03-18 (Actual); Study Completion 2017-03-18 (Actual)

PRIMARY OUTCOMES:
5km - Cycling Time Trial | 2hour
  Time to completion 5 km cycling time trial in the heat

SECONDARY OUTCOMES:
Rectal Temperature | 2hour
  Body core temperature at the end of the 5 km time trial

CONTACTS AND LOCATIONS:
Overall Officials: Stavros A Kavouras, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas - HPER, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No